CLINICAL TRIAL: NCT03514303
Title: Microassay and Allergy Skin Prick Test Correlation Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: United Allergy Services (Industry)
Responsible Party: Sponsor
Other Study IDs: Microassay study-1
Record Dates: First submitted 2018-01-25; First posted 2018-05-02 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-01

CONDITIONS: Allergy Pollen
Keywords: Skin test, Microarray test
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Subject or sub-investigator will perform the finger prick and blot using the instructions listed on the Allergenex sample collection packet. The sample will be mailed to Spiriplex to be analyzed using their microarray device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (10):
- Ragweed: Subjects will test positive or negative to the allergen Ragweed.
  Interventions: Diagnostic Test: Spiriplex Allergenex Microassay
- Timothy Grass: Subjects will test positive or negative to the allergen Timothy Grass.
  Interventions: Diagnostic Test: Spiriplex Allergenex Microassay
- Johnson Grass: Subjects will test positive or negative to the allergen Johnson Grass.
  Interventions: Diagnostic Test: Spiriplex Allergenex Microassay
- Bermuda Grass: Subjects will test positive or negative to the allergen Bermuda Grass.
  Interventions: Diagnostic Test: Spiriplex Allergenex Microassay
- Cladosporium: Subjects will test positive or negative to the allergen Cladosporium.
  Interventions: Diagnostic Test: Spiriplex Allergenex Microassay
- Cat Dander: Subjects will test positive or negative to the allergen Cat Dander.
  Interventions: Diagnostic Test: Spiriplex Allergenex Microassay
- Cockroach: Subjects will test positive or negative to the allergen Cockroach.
  Interventions: Diagnostic Test: Spiriplex Allergenex Microassay
- Dust Mite: Subjects will test positive or negative to the allergen Dust Mite.
  Interventions: Diagnostic Test: Spiriplex Allergenex Microassay
- Oak: Subjects will test positive or negative to the allergen Oak.
  Interventions: Diagnostic Test: Spiriplex Allergenex Microassay
- Dog Dander: Subjects will test positive or negative to the allergen Dog Dander.
  Interventions: Diagnostic Test: Spiriplex Allergenex Microassay

INTERVENTIONS:
Diagnostic Test: Spiriplex Allergenex Microassay — A microassay test using a minimal blood draw for purposes of testing the allergenicity of a subject to specific allergenic proteins.

SUMMARY:
The purpose of this study is to evaluate the potential correlation of the results of allergen-specific skin prick tests (SPT) to that of allergen-specific microarray determination (microassay test). Subjects who meet enrollment criteria, after signing an IRB approved consent form, will perform a minor finger prick blood draw and blot to be mailed off for microassay analysis. Specific statistical analysis will be done to assess all potential correlations between SPT and microassay. This study design should enable assessment of the level of correlation between SPT results and microassay results for specified allergens within a cohort of subjects with allergic rhinitis.

DETAILED DESCRIPTION:
Prospective subjects for study entry will initially be screened by the results of their allergy skin test that were acquired within the past two years. In order to be a prospective subject positive SPT results of five of the following ten allergens will be required: Dust Mite, Ragweed, Cat Dander, Johnson Grass, Bermuda Grass, Timothy Grass, Oak, Cladosporium, Dog Dander, and Cockroach. After signing an IRB approved consent form, these patients will undergo a finger prick blood draw and blot. This study will be conducted in compliance with the protocol, GCP and applicable regulatory requirements.

Subjects 18 years of age or over who have never initiated a course of allergy immunotherapy or have not completed more than three months of SCIT immunotherapy will be enrolled.

Sub-investigator(s) will screen patient charts from a database of patients previously tested using the UAS protocol. Patients that qualify based on inclusion criteria will be contacted by phone and asked if they would be willing to participate in this study.

Subject arrives to the clinic and all inclusion and exclusion criteria are verified by their primary physician and the sub-investigator. Sub-investigator insures that the IRB verified consent form is signed and that the patient has no questions. Subject or sub-investigator will perform the finger prick and blot using the instructions listed on the Allergenex sample collection packet. The sample will be mailed to Spiriplex to be analyzed using their microarray device. The microassay results will be sent to the primary investigation site for correlation analysis with the previously logged SPT results. These results will be blinded to the statisticians and researchers that will be determining potential correlation between SPT and microassay results.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years of age or over who have never initiated a course of allergy immunotherapy or have not completed more than three months of subcutaneous immunotherapy will be enrolled.

Exclusion Criteria:

* Subjects with bleeding disorders or a history of vasovagal reactions to blood draws will not be enrolled in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects 18 years of age or over who have never initiated a course of allergy immunotherapy or have not completed more than three months of subcutaneous immunotherapy will be enrolled. They will have performed an allergen specific skin prick test within the last 2 years through United Allergy Services.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Microassay Tests Completion | 2-3 months
  All patients will be tested by microassay for the 10 allergen groups for comparison to historic skin prick tests of the same 10 allergens.

CONTACTS AND LOCATIONS:
Locations (1):
- United Allergy Services, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No